CLINICAL TRIAL: NCT02280161
Title: An Investigation of the Role of Germ-Line Mutations in Cancer Predisposition, Tumor Biology, and Response to Treatment
Brief Title: Germ-Line Mutations in Blood and Saliva Samples From Patients With Cancer
Status: Recruiting | Type: Observational
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 14-001115; NCI-2014-02065 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); JCCCID488 (Other: Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A blood sample of 30mL or a saliva collection (obtained by spitting into a special collection cup) will be obtained from each patient.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (germ-line mutation analysis): Patients undergo collection of blood and saliva samples 1-3 times at the discretion of the investigator for germ-line mutation analysis.
  Interventions: Other: cytology specimen collection procedure

INTERVENTIONS:
Other: cytology specimen collection procedure — Correlative studies
  Other Names: cytologic sampling

SUMMARY:
This research trial studies germ-line mutations in blood and saliva samples from patients with cancer. Studying samples of blood and saliva from patients with cancer in the laboratory may help doctors learn more about how inherited genetic mutations can affect cancer predisposition (an inherited increase in the risk of developing cancer), their impact on treatment response, and their role in cancer development.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To collect germ-line deoxyribonucleic acid (DNA) and nucleic acids from cancer patients to further investigate the association and identify new germ-line mutations that impact cancer predisposition.

II. To investigate the role of germ-line mutations in predicting cancer outcome and response to therapy.

SECONDARY OBJECTIVES:

I. To determine the effect of the identified variants on tumor micro-ribonucleic acid (miRNA), protein and gene expression.

II. To study expression of DNA, ribonucleic acid (RNA) or protein in the blood of cancer patients with and without variants of interest to discover correlations between such levels and the presence of cancer and/or response to therapy in these patients.

OUTLINE:

Patients undergo collection of blood and saliva samples 1-3 times at the discretion of the investigator for germ-line mutation analysis.

After completion of study, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or clinical confirmed tissue diagnosis of a cancer
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients will be excluded if their cancer cannot be confirmed
* Refusal to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a confirmed diagnosis of cancer.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-09-16 (Actual); Primary Completion 2026-09-16 (Estimated); Study Completion 2027-09-16 (Estimated)

PRIMARY OUTCOMES:
Prevalence of germ-line variants | Up to 5 years
  The prevalence of germ-line variants of interest will be compared to the baseline prevalence found using available large human genomic DNA collections. The primary statistical analysis will involve comparisons of genotypes between with (cases) and without (controls) the germ-line mutation. This analysis will include Pearson's chi-square analysis or Fisher's exact test and computation of odds ratios to assess the relationship of the genetic polymorphism and cancer risk.
Overall genotype frequencies | Up to 5 years
  The overall genotype frequencies among the cases and expected control levels will first be compared with the frequencies expected from Hardy-Weinberg equilibrium by goodness-of-fit chi-square. Odds ratios and 95% confidence intervals will be used to estimate risk associated with the variant genotypes by using both univariate and unconditional multivariate logistic regression models.
Response to treatment | Up to 5 years
  The impact of inherited variants on response to treatment will be determined.
Cancer development | Up to 5 years
  The role of inherited variants in clinical and pathological cancer development will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Weidhaas, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, Los Angeles, California, United States